CLINICAL TRIAL: NCT05783726
Title: Testing Product Messages in Colombia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Universidad Nacional de Colombia (Other); The Bloomberg Family Foundation, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-0401b
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Other): The control arm will show the products with no label.
  Interventions: Other: Control
- Experimental: Nutriscore Label (Experimental): The Nutriscore label applies a letter grade (A, B, C, D or E) to a product based on certain nutrient criteria.
  Interventions: Behavioral: Nutriscore Label
- Experimental: Adapted Peruvian Nutrient Label (Experimental): The adapted label is a black octagon with the words in Spanish saying "Excess of sugar,"Excess of saturated fat," or "Excess of salt/sodium" depending on the nutrition contents of the product. Below the octagon is a box with words in Spanish saying "Avoid high consumption"
  Interventions: Behavioral: Adapted Peruvian Nutrient Label
- Experimental: Guideline Daily Amount Label (Experimental): The Guideline Daily Amount label highlights the nutrient contents of the product by serving. It lists the calories, total fat, saturated fat, sugar, and sodium, as well are their % of the daily value.
  Interventions: Behavioral: Guideline Daily Amount Label

INTERVENTIONS:
Other: Control — Participants will be shown images of juice, bread, yogurt, cookies, and cereal without any added front-of-package labels.
  Arms: Control
Behavioral: Nutriscore Label — A front-of-package Nutriscore label will be applied to images of juice, bread, yogurt, cookies, and cereal. This label applies a score of A, B, C, D, or E based on the product's nutrition profile.
  Arms: Experimental: Nutriscore Label
Behavioral: Adapted Peruvian Nutrient Label — A front-of-package octagonal nutrient label will be applied to images of juice, bread, yogurt, cookies, and cereal. The label text informs consumers if a product is high in sugar, saturated fat, or salt/sodium. These labels were developed by the Peruvian government and adapted by investigators.
  Arms: Experimental: Adapted Peruvian Nutrient Label
Behavioral: Guideline Daily Amount Label — A front-of-package Guideline Daily Amount label will be applied to images of juice, bread, yogurt, cookies, and cereal. The label shows the amount and percent of daily value of calories, total fat, saturated fat, sugar, and sodium in one serving of a product.
  Arms: Experimental: Guideline Daily Amount Label

SUMMARY:
Purpose: To better understand the impact of different front-of-package labels (FOPLs) on consumer purchasing intentions and ability to identify unhealthy foods.

Participants: ~8,000 Colombians, recruited from Offerwise, that are 18 years or older.

Procedures (methods): Participants will be randomly assigned to view images of food and drink products with either a nutrient warning label, Guideline Daily Amount label, Nutriscore label, or no-label control. They will be asked a series of questions about the products and the labels (excluding control group) on them. Questions will also include standard demographic and health related variables.

DETAILED DESCRIPTION:
Participants will be recruited from Offerwise (an online panel research company). Following online consent, participants will be randomly assigned to view different labels (explained below) on food and drink packaging. Participants will answer self-reported responses to the content (e.g., elaboration, beliefs, perceived healthfulness). After being randomized to one of the four groups and answering questions (e.g. which product is healthier, which product would you buy), the participant will see all three labels and select which is most dissuading from consuming a product high in a nutrient. At the end, the participant will answer demographic questions.

Participants will be randomized to see either a no-label control or 1 of 3 nutrient labels. The participants will see 5 types of products with the labels (fruit drinks, yogurt, sliced bread, cookies, and breakfast cereal).

Nutrient labels:

1. Guideline Daily Amount label
2. Nutriscore label
3. Adapted Peruvian nutrient warning label (high in sugar, high in saturated fat, high in salt/sodium)

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old
* Resident of Colombia
* Offerwise panel member (recruitment platform)

Exclusion Criteria:

* <18 years old or >64 years old
* Not a resident of Colombia

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8086 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Selection of Product Higher in Sugar | During ~15 minute online survey
  Percentage of participants who select the less healthy product in a set of two products as the product the consumer most wants to buy.
Correct Identification of the Product Higher in Sugar | During ~15 minute online survey
  Percentage of participants who correctly select the product higher in sugar (between two products)

SECONDARY OUTCOMES:
Perceived Message Effectiveness | During ~15 minute online survey
  Perceived message effectiveness of the study labels. Response options are on a 1 to 5 scale, with lower scores representing a higher amount of the construct.
  Perceived message effectiveness is measured using 3 items adapted from Baig et al. (2018): concern, unpleasantness, and discouragement. Responses to the 3 items will be averaged to create a perceived message effectiveness score.
  Question: How much does this message...
  make you concerned about the health effect of consuming an unhealthy product? discourage you from wanting to eat an unhealthy product? make eating an unhealthy product seem unpleasant to you? Only asked of the label arms, not control.
Purchase Likelihood | During ~15 minute online survey
  Likelihood that participants would purchase this product in the next week if it were available. Response options are on a 1 to 5 scale, with lower scores representing a higher amount of the construct
Identify Less Healthy Product | During ~15 minute online survey
  Percentage of participants that correctly identify the less healthy product when selecting between two products.
Ability to Identify Product as Having Excess of Sugar/Saturated Fat/Sodium | During ~15 minute online survey
  Percentage of participants who correctly identify that the product contains excess sugar, saturated fat, or sodium.
Most Discouraging Label | During ~15 minute online survey
  Percentage of participants selecting each nutrient label as most discouraging them from consuming the product.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey S Taillie, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Carolina Population Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mora-Plazas M, Higgins ICA, Gomez LF, Hall MG, Parra MF, Bercholz M, Murukutla N, Taillie LS. Impact of nutrient warning labels on Colombian consumers' selection and identification of food and drinks high in sugar, sodium, and saturated fat: A randomized controlled trial. PLoS One. 2024 Jun 10;19(6):e0303514. doi: 10.1371/journal.pone.0303514. eCollection 2024. PMID 38857209

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/26/NCT05783726/Prot_SAP_ICF_001.pdf